CLINICAL TRIAL: NCT05344495
Title: Efficacy of Median Nerve Hydrodissection by Hyalase Versus Midazolam in the Treatment of Carpal Tunnel Syndrome: A Randomized, Clinical Trial.
Brief Title: Efficacy of Median Nerve Hydrodissection by Hyalase Versus Midazolam in the Treatment of Carpal Tunnel Syndrome:
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mina Maher, Lecturer of anesthesia and ICU, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 277/4-2022
Record Dates: First submitted 2022-04-14; First posted 2022-04-25 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Pain, Neuropathic
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hyalse group (Active Comparator): ultrasonographic median nerve hydrodissection by hyalase and bupivacaine 0.5%
  Interventions: Drug: hyalase group
- midazolam group (Active Comparator): ultrasonographic median nerve hydrodissection by midazolam and bupivacaine 0.5%
  Interventions: Drug: midazolam group

INTERVENTIONS:
Drug: hyalase group — bupivacaine 15 mg 0.5% plus 2 mL normal saline containing 300 international units (IU) hyaluronidase.
  Other Names: Sonar guided median nerve hydrodissection by hyalase and bupivacaine 0.5%
  Arms: hyalse group
Drug: midazolam group — 2 mg midazolam dissolved in 2 ml sterile saline plus 15 mg bupivacaine 0.5%
  Other Names: Sonar guided median nerve hydrodissection by midazolam and bupivacaine 0.5%
  Arms: midazolam group

SUMMARY:
Comparing efficacy of hyalase and midazolam in median nerve entrapement neuropathy

ELIGIBILITY:
Inclusion Criteria:

* adult patients (30 - 70 years old) complaining of carpal tunnel syndrome of 3 month duration or more , diagnosed axonal neuropathy using electrodiagnosis , nerve conduction study refractory to medical treatment for 2 months .

Exclusion Criteria:

* Diabetic patients
* Pregnant population .
* Refusal to participate

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-07-20 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
pain score | 6 months
  visual analogue score which represents 0 = no pain, 10= worst un-imaginable pain

SECONDARY OUTCOMES:
Boston questionnaire | 6 months
  symptom severity ... function severity
median nerve sonogrphy | 6 months
  cross sectional area
Nerve electrophysiology | 6 months
  sensory velocity and distal motor latency ... 1m/sec is the least and 10m/sec is the highest

CONTACTS AND LOCATIONS:
Locations (1):
- Mina Raouf, ALMinya, Minya Governorate, Egypt